CLINICAL TRIAL: NCT03408704
Title: The Effectiveness of an Antimicrobial Stewardship Program (ASP) in Primary Health Care in the Management of Patients With a Sore Throat
Brief Title: Antimicrobial Stewardship Program (ASP) in Patients With a Sore Throat
Acronym: ASP-Throat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: James Cook University, Queensland, Australia (Other); Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: U1111-1207-9573
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-02

CONDITIONS: Tonsillitis; Streptococcus Pharyngitis; Sore Throat; Pharyngitis; Pharyngitis Bacterial
Keywords: Streptococcus Pyogenes Infection; Randomized Controlled Trial
MeSH Terms: conditions — Tonsillitis; Pharyngitis; Streptococcal Infections

STUDY DESIGN:
Intervention Model Description: Parallel group randomized controlled trial. Primary health care clinics are randomized. The enrolment number refers to included clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASP-arm (Experimental): This group of primary health care centers get the internal education (ASP).
  Interventions: Other: ASP
- Control-arm (No Intervention): No intervention at all.

INTERVENTIONS:
Other: ASP — It consists of one educational session where doctors and staff at the center discuss current guidelines around management of patients attending for a sore throat. At the education the following is discussed:
  1. The Swedish guidelines
  2. Example of cases
  3. Statistics from previous 6 month showing how well this clinic adheres to the Swedish guidelines.
  Arms: ASP-arm

SUMMARY:
The investigators have developed an antibiotic stewardship program (ASP) to increase adherence to the Swedish guidelines for managing patients with a sore throat. This is a randomized controlled trial where primary health care centers are randomised to get the ASP or not. The adherence to the Swedish guidelines are measured in all participating centers.

DETAILED DESCRIPTION:
The investigators have developed an antibiotic stewardship program (ASP) to increase adherence to the Swedish guidelines for managing patients with a sore throat. This is a randomized controlled trial where primary health care centers are randomised to get the ASP or not. The adherence to the Swedish guidelines are measured in all participating centers 6 months before and after implementation of the ASP. The ASP consists of educational meetings at the clinic for medical practitioners and nurses being informed about current guidelines, seeing their clinics adherence to the guidelines as well as discussing cases.

ELIGIBILITY:
Inclusion Criteria:

* Being a primary health care center in the Vastra Gotaland region, Sweden accepting participation

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The effect of an ASP on the change in proportion of positive RADT among patients prescribed AB - 6m | Pre intervention 6 Months period compared to the 6 months period prior to follow-up at 6 months
  The effect of an antibiotic stewardship program (ASP) on the proportion of patients prescribed antibiotics (J01 excluding methenamine) for a sore throat where a rapid antigen detection test (RADT) to detect Group A Streptococcus (GAS) is taken and is positive. Change from a 6 month period before initiation of the intervention (baseline) is compared with a time period of 6 months prior to the follow up date.
  The change from baseline to follow-up in all primary health care centres (PHCC) in the intervention group is compared to the corresponding change in PHCC in the control group (ASP group versus control group) using linear regression where adjustment will also be made for: the number of enlisted patients at baseline, location in cities versus small villages, Adjusted Clinical Group (ACG), Care-need index (CNI) and type of PHCC (private/public).
The effect of an ASP on the change in proportion of positive RADT among patients prescribed AB - 12m | Pre intervention 6 Months period compared to the 6 months period prior to follow-up at 12 months
  The effect of an antibiotic stewardship program (ASP) on the proportion of patients prescribed antibiotics (J01 excluding methenamine) for a sore throat where a rapid antigen detection test (RADT) to detect Group A Streptococcus (GAS) is taken and is positive. Change from a 6 month period before initiation of the intervention (baseline) is compared with a time period of 6 months prior to the follow up date.
  The change from baseline to follow-up in all primary health care centres (PHCC) in the intervention group is compared to the corresponding change in PHCC in the control group (ASP group versus control group) using linear regression where adjustment will also be made for: the number of enlisted patients at baseline, location in cities versus small villages, Adjusted Clinical Group (ACG), Care-need index (CNI) and type of PHCC (private/public).
The effect of an ASP on the change in proportion of positive RADT among patients prescribed AB - 18m | Pre intervention 6 Months period compared to the 6 months period prior to follow-up at 18 months
  The effect of an antibiotic stewardship program (ASP) on the proportion of patients prescribed antibiotics (J01 excluding methenamine) for a sore throat where a rapid antigen detection test (RADT) to detect Group A Streptococcus (GAS) is taken and is positive. Change from a 6 month period before initiation of the intervention (baseline) is compared with a time period of 6 months prior to the follow up date.
  The change from baseline to follow-up in all primary health care centres (PHCC) in the intervention group is compared to the corresponding change in PHCC in the control group (ASP group versus control group) using linear regression where adjustment will also be made for: the number of enlisted patients at baseline, location in cities versus small villages, Adjusted Clinical Group (ACG), Care-need index (CNI) and type of PHCC (private/public).

SECONDARY OUTCOMES:
The effect of an ASP on the change in proportion of negative RADT given AB - 6m | Pre intervention 6 Months period compared to the 6 months period prior to follow-up at 6 months
  The effect of an antibiotic stewardship program (ASP) on the proportion of patients prescribed antibiotics (J01 excluding methenamine) for a sore throat where a rapid antigen detection test (RADT) to detect Group A Streptococcus (GAS) is taken and is negative being. Change from a 6 month period before initiation of the intervention (baseline) is compared with a time period of 6 months prior to the follow up date.
  The change from baseline to follow-up in all primary health care centres (PHCC) in the intervention group is compared to the corresponding change in PHCC in the control group (ASP group versus control group) using linear regression where adjustment will also be made for: the number of enlisted patients at baseline, location in cities versus small villages, Adjusted Clinical Group (ACG), Care-need index (CNI) and type of PHCC (private/public).
The effect of an ASP on the change in proportion of negative RADT given AB - 12m | Pre intervention 6 Months period compared to the 6 months period prior to follow-up at 12 months
  The effect of an antibiotic stewardship program (ASP) on the proportion of patients prescribed antibiotics (J01 excluding methenamine) for a sore throat where a rapid antigen detection test (RADT) to detect Group A Streptococcus (GAS) is taken and is negative being. Change from a 6 month period before initiation of the intervention (baseline) is compared with a time period of 6 months prior to the follow up date.
  The change from baseline to follow-up in all primary health care centres (PHCC) in the intervention group is compared to the corresponding change in PHCC in the control group (ASP group versus control group) using linear regression where adjustment will also be made for: the number of enlisted patients at baseline, location in cities versus small villages, Adjusted Clinical Group (ACG), Care-need index (CNI) and type of PHCC (private/public).
The effect of an ASP on the change in proportion of negative RADT given AB - 18m | Pre intervention 6 Months period compared to the 6 months period prior to follow-up at 18 months
  The effect of an antibiotic stewardship program (ASP) on the proportion of patients prescribed antibiotics (J01 excluding methenamine) for a sore throat where a rapid antigen detection test (RADT) to detect Group A Streptococcus (GAS) is taken and is negative being. Change from a 6 month period before initiation of the intervention (baseline) is compared with a time period of 6 months prior to the follow up date.
  The change from baseline to follow-up in all primary health care centres (PHCC) in the intervention group is compared to the corresponding change in PHCC in the control group (ASP group versus control group) using linear regression where adjustment will also be made for: the number of enlisted patients at baseline, location in cities versus small villages, Adjusted Clinical Group (ACG), Care-need index (CNI) and type of PHCC (private/public).
The effect of an ASP on the change in proportion of recommended AB prescribed - 6m | Pre intervention 6 Months period compared to the 6 months period prior to follow-up at 6 months
  The effect of an antibiotic stewardship program (ASP) on the proportion of patients prescribed PcV compared to all patients prescribed any antibiotics (J01 excluding methenamine) for a sore throat. Change from a 6 month period before initiation of the intervention (baseline) is compared with a time period of 6 months prior to the follow up date.
  The change from baseline to follow-up in all primary health care centres (PHCC) in the intervention group is compared to the corresponding change in PHCC in the control group (ASP group versus control group) using linear regression where adjustment will also be made for: the number of enlisted patients at baseline, location in cities versus small villages, Adjusted Clinical Group (ACG), Care-need index (CNI) and type of PHCC (private/public).
The effect of an ASP on the change in proportion of recommended AB prescribed - 12m | Pre intervention 6 Months period compared to the 6 months period prior to follow-up at 12 months
  The effect of an antibiotic stewardship program (ASP) on the proportion of patients prescribed PcV compared to all patients prescribed any antibiotics (J01 excluding methenamine) for a sore throat. Change from a 6 month period before initiation of the intervention (baseline) is compared with a time period of 6 months prior to the follow up date.
  The change from baseline to follow-up in all primary health care centres (PHCC) in the intervention group is compared to the corresponding change in PHCC in the control group (ASP group versus control group) using linear regression where adjustment will also be made for: the number of enlisted patients at baseline, location in cities versus small villages, Adjusted Clinical Group (ACG), Care-need index (CNI) and type of PHCC (private/public).
The effect of an ASP on the change in proportion of recommended AB prescribed - 18m | Pre intervention 6 Months period compared to the 6 months period prior to follow-up at 18 months
  The effect of an antibiotic stewardship program (ASP) on the proportion of patients prescribed PcV compared to all patients prescribed any antibiotics (J01 excluding methenamine) for a sore throat. Change from a 6 month period before initiation of the intervention (baseline) is compared with a time period of 6 months prior to the follow up date.
  The change from baseline to follow-up in all primary health care centres (PHCC) in the intervention group is compared to the corresponding change in PHCC in the control group (ASP group versus control group) using linear regression where adjustment will also be made for: the number of enlisted patients at baseline, location in cities versus small villages, Adjusted Clinical Group (ACG), Care-need index (CNI) and type of PHCC (private/public).
The effect of an ASP on the change in proportion of patients where CRP is requested - 6m | Pre intervention 6 Months period compared to the 6 months period prior to follow-up at 6 months
  The effect of an antibiotic stewardship program (ASP) on the proportion of patients diagnosed with pharyngotonsillitis where the lab test C-reactive protein (CRP) is requested. Change from a 6 month period before initiation of the intervention (baseline) is compared with a time period of 6 months prior to the follow up date.
  The change from baseline to follow-up in all primary health care centres (PHCC) in the intervention group is compared to the corresponding change in PHCC in the control group (ASP group versus control group) using linear regression where adjustment will also be made for: the number of enlisted patients at baseline, location in cities versus small villages, Adjusted Clinical Group (ACG), Care-need index (CNI) and type of PHCC (private/public).
The effect of an ASP on the change in proportion of patients where CRP is requested - 12m | Pre intervention 6 Months period compared to the 6 months period prior to follow-up at 12 months
  The effect of an antibiotic stewardship program (ASP) on the proportion of patients diagnosed with pharyngotonsillitis where the lab test C-reactive protein (CRP) is requested. Change from a 6 month period before initiation of the intervention (baseline) is compared with a time period of 6 months prior to the follow up date.
  The change from baseline to follow-up in all primary health care centres (PHCC) in the intervention group is compared to the corresponding change in PHCC in the control group (ASP group versus control group) using linear regression where adjustment will also be made for: the number of enlisted patients at baseline, location in cities versus small villages, Adjusted Clinical Group (ACG), Care-need index (CNI) and type of PHCC (private/public).
The effect of an ASP on the change in proportion of patients where CRP is requested - 18m | Pre intervention 6 Months period compared to the 6 months period prior to follow-up at 18 months
  The effect of an antibiotic stewardship program (ASP) on the proportion of patients diagnosed with pharyngotonsillitis where the lab test C-reactive protein (CRP) is requested. Change from a 6 month period before initiation of the intervention (baseline) is compared with a time period of 6 months prior to the follow up date.
  The change from baseline to follow-up in all primary health care centres (PHCC) in the intervention group is compared to the corresponding change in PHCC in the control group (ASP group versus control group) using linear regression where adjustment will also be made for: the number of enlisted patients at baseline, location in cities versus small villages, Adjusted Clinical Group (ACG), Care-need index (CNI) and type of PHCC (private/public).
Proportion of patients given AB for a sore throat with no throat swab taken | Pre intervention 6 Months period
  The proportion of patients given a diagnosis of pharyngotonsillitis and prescribed AB (J01 excluding methenamine) where a throat swab is not taken.
  Descriptive statistics is presented and a group comparison is not made.
Proportion of patients with pharyngotonsillitis where a throat swab is taken and sent for a culture | Pre intervention 6 Months period
  The proportion of patients given a diagnosis of pharyngotonsillitis and where a throat swab is taken and send to a microbiologic laboratory for a throat culture.
  Descriptive statistics is presented and a group comparison is not made.
Proportion of patients with pharyngotonsillitis where a test for mononucleosis is taken | Pre intervention 6 Months period
  The proportion of patients given a diagnosis of pharyngotonsillitis and where a test for mononucleosis is taken.
  Descriptive statistics is presented and a group comparison is not made.

CONTACTS AND LOCATIONS:
Overall Officials: Pär-Daniel Sundvall, MD PhD, Principal Investigator — Vastra Gotaland region, Sweden
Locations (1):
- vastra Gotaland region, Borås, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No
The data will be summary data for each participating primary health care clinic. The investigators will publish the summary of all clinics but don't intend to show data from single clinics.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT03408704/Prot_SAP_000.pdf